CLINICAL TRIAL: NCT07387588
Title: Anemia as Predictor of Outcome in IBD Pateints in Assuit University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa Kotb Abdullah Hassan, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: Anemia IDB
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Adult patients (≥18 years old) diagnosed with inflammatory bowel diseases (ulcerative colitis or Crohn's disease).

SUMMARY:
Inflammatory bowel diseases (IBD), encompassing ulcerative colitis (UC) and Crohn's disease (CD), are chronic, relapsing inflammatory disorders of the gastrointestinal tract with significant morbidity and impact on patients' quality of life. Despite advances in diagnostic and therapeutic strategies, many patients continue to experience complications, frequent hospitalizations, and impaired long-term outcomes. Identifying prognostic factors that can predict disease course and response to therapy is therefore crucial in guiding clinical management and optimizing resource utilization.

Anemia is one of the most frequent extraintestinal manifestations of IBD, with prevalence estimates ranging from 20% to 70% depending on disease activity and population studied. The pathogenesis of anemia in IBD is multifactorial, including iron deficiency due to chronic intestinal blood loss, anemia of chronic disease driven by inflammation, vitamin B12 or folate deficiency, and medication-related bone marrow suppression. Anemia has been consistently associated with increased disease activity, reduced health-related quality of life, higher rates of hospitalization, and poorer overall prognosis in IBD patients.

Given its potential as a simple and accessible biomarker, hemoglobin level and anemia status may serve as valuable predictors of disease outcome. However, local data from Egyptian populations, particularly from Assiut University Hospitals, remain scarce. Studying anemia as a prognostic factor in IBD patients may provide insight into disease severity, help stratify patients at higher risk, and support the development of tailored therapeutic and monitoring strategies. This research aims to fill this knowledge gap by evaluating the prognostic significance of anemia in IBD patients managed at Assiut University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (≥18 years old) diagnosed with inflammatory bowel diseases (ulcerative colitis or Crohn's disease).

  * Patients admitted or followed up in Assiut University Hospitals during the study period.
  * Patients who have given written informed consent to participate in the study.

Exclusion Criteria:

* • Patients with other chronic hematological disorders unrelated to IBD (e.g., aplastic anemia, hemoglobinopathies).

  * Patients with concurrent chronic renal failure, liver failure, or other systemic diseases causing anemia.
  * Patients receiving recent blood transfusion (within the last 3 months) before enrollment
  * Pregnant or lactating women.
  * Patients unwilling or unable to complete the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) diagnosed with inflammatory bowel diseases (ulcerative colitis or Crohn's disease).
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
hospitalization rate | baseline